CLINICAL TRIAL: NCT07179445
Title: A Retrospective Study of Deoxyribonucleic Acid and Ribonucleic Acid Next-Generation Sequencing in Non-Small Cell Lung Cancer Patients With Non-Pathologic Complete Response Following Neoadjuvant Immunotherapy
Brief Title: Analysis of Deoxyribonucleic Acid and Ribonucleic Acid Next-Generation Sequencing in Non-Small Cell Lung Cancer Patients Without Pathological Complete Response Following Neoadjuvant Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Dongsheng Yue, Chief Physician of Surgery, Tianjin Medical University Cancer Institute and Hospital
Other Study IDs: LUAD-non-pCR-001
Record Dates: First submitted 2025-09-07; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: NSCLC
Keywords: NSCLC; Neoadjuvant; NGS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
This multicenter, retrospective cohort study plans to enroll patients with lung adenocarcinoma who received neoadjuvant immunotherapy prior to surgery and did not achieve pathological complete response (non-pCR) upon postoperative pathological evaluation. Using Deoxyribonucleic Acid(DNA) and Ribonucleic Acid(RNA) next-generation sequencing (NGS), the investigators aim to detect driver genetic alterations to investigate the real-world frequency of driver gene positivity in postoperative samples from patients with lung adenocarcinoma-whose EGFR and ALK status had been previously excluded via pathological complete response(pCR) or DNA-based next-generation sequencing-yet still did not attain pathological complete response(pCR) after neoadjuvant immunotherapy. Additionally, the study will characterize the driver-positive patient subgroup and compare the efficacy of postoperative adjuvant immunotherapy between driver-positive and driver-negative populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, regardless of sex.
* Pathologically confirmed, resectable non-small cell lung cancer (NSCLC); having received neoadjuvant therapy containing immune checkpoint inhibitors prior to surgery; without achieving pathological complete response (non-pCR) upon postoperative pathological assessment.
* Molecular characteristics: Pre-treatment biopsy specimens tested negative for EGFR mutations and ALK fusions by DNA-based NGS or PCR methods.
* Sample requirements: Availability of 5-10 formalin-fixed, paraffin-embedded (FFPE) sections prepared from surgical tissue specimens, with ≥5% tumor cell content confirmed by H&E staining.

Exclusion Criteria:

* Failure to meet any one of the requisite eligibility criteria specified in the inclusion criteria.
* History of a concurrent or prior malignancy at other sites.
* Failure to complete the planned cycles of neoadjuvant immunotherapy due to treatment-related toxicities.
* Any other condition that, in the judgment of the investigator, renders the patient unsuitable for participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter, retrospective cohort study plans to enroll patients with non-small cell lung cancer (NSCLC). Cases meeting the eligibility criteria between January 2022 and December 2024 will first be identified through the hospital pathology information management system. The screening process consists of two stages:
  Initial Screening: Extraction of data from electronic medical records for patients aged ≥18 years, with pathologically confirmed NSCLC, and who underwent genetic testing prior to surgery.
  Collection of Neoadjuvant Immunotherapy Information:
  1. Received preoperative neoadjuvant immunotherapy, including regimens such as immune monotherapy, immune combination chemotherapy, or immune combination with antiangiogenic agents, with available postoperative pathological assessment results;
  2. Exclusion of EGFR and ALK positivity in pre-treatment biopsy samples;
  3. Availability of qualifying surgical tissue samples. Estimating a requirement of 300 cases.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of driver-alteration-positive patients detected by combined DNA+RNA testing | through study completion, an average of 1 year
  We selected patients with lung adenocarcinoma who had received preoperative neoadjuvant immunotherapy, did not achieve pathological complete response (pCR) after surgery, and had pre-treatment biopsy samples testing negative for EGFR and ALK alterations. Subsequent combined DNA/RNA next-generation sequencing (NGS) was performed using the 3DMed Onco™ Core Tissue Detection Kit. The proportion of patients with identified driver genomic alterations served as the primary endpoint of the study.

SECONDARY OUTCOMES:
Comparative Analysis of Adjuvant Immunotherapy Efficacy Between Driver-Alteration-Positive and Negative Cohorts | through study completion, an average of 1 year
  For the comparison between driver gene-positive and negative populations:
  Disease-Free Survival (DFS) will be compared between patients who received adjuvant immunotherapy and were driver gene-positive versus those who were driver gene-negative. DFS is defined as the time from surgery to the first occurrence of disease recurrence, distant metastasis, or death from any cause.
Stratified Analysis of EGFR/ALK-Positive Versus Other Driver-Alteration-Positive Subgroups | through study completion, an average of 1 year
  For the stratified analysis among positive populations:
  Among the driver gene-positive patients who received adjuvant immunotherapy, a stratified analysis will be performed comparing patients with EGFR or ALK mutations versus those with mutations in other driver genes (e.g., ROS1, BRAF V600E, MET, RET, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital(Lead Center), Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT07179445/Prot_000.pdf